CLINICAL TRIAL: NCT06463691
Title: An Open-label, Multi-center, Single-arm Study to Evaluate the Efficacy and Safety of Sonrotoclax, Zanubrutinib and CD20mab in Untreated MCL Patients
Brief Title: Sonrotoclax, Zanubrutinib and CD20mab in Untreated MCL Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417- 2003-IIT
Record Dates: First submitted 2024-06-05; First posted 2024-06-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: MCL
Keywords: MCL; Sonrotoclax; Zanubrutinib
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Intervention Model Description: Sonrotoclax, Zanubrutinib and CD20mab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Sonrotoclax, orally, 320 mg once daily following ramp-up. Zanubrutinib, orally, 320 mg total daily dose. CD20mab, which is recommended Rituximab, 375mg/m2, from C1 to C12
  Interventions: Drug: BGB-11417; Drug: BGB-3111; Drug: CD20

INTERVENTIONS:
Drug: BGB-11417 — Sonrotoclax, orally, 320 mg once daily following a weekly ramp-up schedule
  Other Names: Sonrtotoclax
Drug: BGB-3111 — Zanubrutinib, orally, 320 mg total daily dose
  Other Names: Zanubrutinib
Drug: CD20 — CD20mab is recommened as Rituximab as per the protocol, other CD20mab is also allowed.

SUMMARY:
This is a an open-label, multi-center, single-arm study to evaluate the efficacy and safety of sonrotoclax, zanubrutinib and CD20mab in untreated MCL patients.

DETAILED DESCRIPTION:
The benefits of efficacy and survival of immunotherapy regimen in TN MCL is limited, and not all patients are fit for receiving chemotherapy. Considering the balance of toxicity and efficacy, a chemo-free regimen will be a trend in 1L MCL patients. The study is to explore the sonrotoclax, zanubrutinib and CD20mab combination regimen for TN MCL.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be ≥ 18 years of age.
2. Subject must have a confirmed Mantle Cell Lymphoma (MCL) diagnosis according to WHO (2008) criteria.
3. Previously untreated MCL
4. Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2.
5. Nonsterile men and women of child-bearing potential must agree to use highly effective contraceptives (e.g., condoms, implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence, or sterilized partner) while on study; this should be maintained for 90 days after the last dose of study drug.
6. Subject must have adequate bone marrow function at Screening as follows:

   a.Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L (neutropenia due to marrow infiltration may be supported by growth factors);

   • b. Platelets ≥ 75,000/mm3 (or ≥ 50,000/mm3 for patients with bone marrow involvement of lymphoma) within 7 days
7. Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening as follows:

   1. aPTT and PT not to exceed 1.5 × the upper limit of normal (ULN); Serum creatinine not to exceed 2 x ULN, and a calculated creatinine clearance of at least 50 mL/min using the Cockcroft-Gault equation or a 24-hour urine collection;
   2. AST or ALT ≤ 3.0 × the upper normal limit (ULN) of institution's normal range; Bilirubin ≤ 1.5 × ULN. Subjects with documented Gilbert's Syndrome may have a bilirubin > 1.5 × ULN.
8. Written informed consent form according to GCP and national regulations.

Exclusion Criteria:

1. Subject has known central nervous system involvement by MCL.
2. Prior malignancy other than MCL within the past 3 years, except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 prostate cancer.
3. Receiving any treatment with a moderate CYP3A4 inhibitor or strong CYP3A4 inhibitor or inducer within 2 weeks (or 5 half-lives, whichever is longer) before the first dose of study drug or requiring long-term use of strong CYP3A4 inhibitors or inducers.
4. Prior ASCT within the last 3 months; or prior autologous chimeric antigen receptor-T cell therapy within the last 3 months; or prior allogeneic stem cell transplant within the last 6 months or currently has an active graft-vs-host disease requiring the use of immunosuppressants.
5. Major surgery within 4 weeks of screening.
6. Clinically significant cardiovascular disease including the following:

   1. Myocardial infarction within 6 months before screening
   2. Unstable angina within 3 months before screening
   3. New York Heart Association class III or IV congestive heart failure
   4. History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation)
   5. QT interval corrected based on Fridericia's formula (QTcF) > 480 msec.
   6. History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place
   7. Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mmHg and diastolic blood pressure > 105 mmHg at screening.
7. Prior exposure to a BCL2 inhibitor (e.g., venetoclax/ABT-199).
8. Prior exposure to a BTK inhibitor (e.g., ibrutinib, zanubrutinib).
9. History of hypersensitivity to excipient(s) of the sonrotoclax tablet.
10. Patients with unresolved hepatitis B or C infection or known HIV-positive infection：

    1. Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) DNA is undetectable (< 20 IU/mL), and if they are willing to undergo monitoring for HBV reactivation.
    2. Presence of hepatitis C virus (HCV) antibody. Patients with presence of HCV antibody are eligible if HCV RNA is undetectable (< 15 IU/mL), and if they are willing to undergo monitoring for HCV reactivation.
11. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
12. Pregnant or lactating women.
13. History of stroke or intracranial hemorrhage within 6 months before the first dose of study drug.
14. Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of safety or efficacy results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
CR (complete response) rate at cycle 12 by investigator (INV). | From enrollment to the end of treatment at the end of cycle 12 (each cycle is 28 days)
  Complete response rate (CRR) of the study population from the initiation of the first cycle treatment. CRR is defined as the proportion of patients that achieved the best response of CR, determined by INV.

SECONDARY OUTCOMES:
ORR (Overall response rate) | From enrollment to the end of treatment at the end of cycle 36 (each cycle is 28 days)
  ORR is defined as the proportion of patients achieving complete response (CR) or partial response (PR), as determined by INV -PFS defined as time from the date of enrollment to the date of first confirmed disease progression or death due to any cause, whichever occurs first, as determined by INV.
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Overall survival (OS) is defined as the duration from the date of initiation of the first cycle of treatment to the date of death because of any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided